CLINICAL TRIAL: NCT05774054
Title: The Impact of Early Norepinephrine Administration on Outcomes of Patients With Sepsis-induced Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: early noradrenaline in sepsis
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Norepinephrine; Sepsis; Hypotension
MeSH Terms: conditions — Sepsis; Hypotension | interventions — Crystalloid Solutions; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): patients received (30ml /kg) ringer's lactate solution after first presentation then norepinephrine was added when persistent mean arterial pressure (MAP)> 65 mmHg despite adequate fluid resuscitation
  Interventions: Drug: Crystalloid
- B (Active Comparator): patients received ( 30ml /kg) ringer's lactate solution after first presentation combined with norepinephrine infusion (0.05 mic/kg/min)
  Interventions: Drug: noradrenaline

INTERVENTIONS:
Drug: Crystalloid — received (30ml /kg) ringer's lactate solution after first presentation then norepinephrine was added when persistent mean arterial pressure (MAP)> 65 mmHg despite adequate fluid resuscitation
  Other Names: late noradrenaline infusion
  Arms: A
Drug: noradrenaline — received ( 30ml /kg) ringer's lactate solution after first presentation combined with norepinephrine infusion (0.05 mic/kg/min)
  Other Names: early noradrenaline infusion
  Arms: B

SUMMARY:
Septic shock is defined as sepsis with persistent hypotension requiring vasopressors to maintain mean arterial pressure (MAP)≥ 65 mmHg and a serum lactate level of > 2 mmol/L (18 mg/dL) despite sufficient volume resuscitation

. Hypovolemia (both relative and absolute) and reduced vascular tone have a role in determining the severity of hypotension in septic shock

DETAILED DESCRIPTION:
Septic shock is defined as sepsis with persistent hypotension requiring vasopressors to maintain mean arterial pressure (MAP)≥ 65 mmHg and a serum lactate level of > 2 mmol/L (18 mg/dL) despite sufficient volume resuscitation . Hypovolemia (both relative and absolute) and reduced vascular tone have a role in determining the severity of hypotension in septic shock

. When mean arterial pressure (MAP) falls below a specific critical level organ blood flow is physiologically dependent on perfusion pressure. Fluid resuscitation and vasopressors have an influence on hypovolemia and the vascular tone in the early phase, as fluid resuscitation aims to correct hypovolemia and vasopressors-norepinephrine (NE)- as a first-line drug aiming to restore vascular tone to assure organ perfusion

. Norepinephrine is both an alpha1- and beta1-agonist so it is able to increase vascular tone and contractility

. Nevertheless, a large amount of fluids will increase the risk of fluid overload, which is a common complication during septic shock resuscitation

* After the early phase, only fifty percent of patients respond to fluid administration, meaning that fluid treatment cannot boost cardiac output (CO) The current data indicate that the time from the onset of septic shock to the initiation of norepinephrine administration is a significant survival predictor; however, a suggestion for the optimal time to provide norepinephrine support was not explicitly expressed

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged from18 to 65 years old
* had the diagnostic criteria for sepsis as the presence of infection
* systemic manifestations of infection and signs of Hypoperfusion

Exclusion Criteria:

* Acute cerebral vascular event
* Active cardiac conditions
* Valvular heart diseases
* Hypotension suspected to be due to another cause and comorbidities
* Status asthmatics
* Active hemorrhage
* Pregnancy
* Burn injury
* Requirement for immediate surgery
* Advanced-stage cancer
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
the required duration to achieve the target MAP | 24 hours since the diagnosis of sepsis
  time to achieve target mean arterial pressure over or equal to 65 mmHg once the diagnosis of sepsis is confirmed, is the target to stop fluid management.

CONTACTS AND LOCATIONS:
Overall Officials: ghada elbarady, MD, Study Director — tanta university, faculty of medicine
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No